CLINICAL TRIAL: NCT01433094
Title: Study on Psychoeducation Enhancing Results of Adherence in Schizophrenia
Acronym: SPERA-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, donatella rita petretto, Assistant Professor, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIFA FARM892ZXE
Record Dates: First submitted 2011-08-20; First posted 2011-09-13 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Patient Non-Compliance; Schizophrenia and Related Disorders
Keywords: Adherence; Psychoeducation; Pharmacotherapy; Schizophrenia; Family support
MeSH Terms: conditions — Patient Compliance; Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Falloon et al. Psychoeducation Program (Experimental): The intervention aims to improve communication and problem-solving abilities in patients and their families by sessions focused on: assessment of the individual's and the family's strengths, weaknesses, and goals; education about schizophrenia and treatment; communication skills training; problem-solving
  Interventions: Behavioral: Falloon et al. Psychoeducation Program
- Generic Treatment (Active Comparator): The comparator is a treatment with generic informative prospect on the disorders and with the same frequencies as the Intervention. Treatment sessions are provided on a weekly basis for 6 months (1 hour for each session) (groups of about 8-9 persons - patients and caregivers).
  Interventions: Behavioral: Generic Treatment

INTERVENTIONS:
Behavioral: Falloon et al. Psychoeducation Program — The intervention aims to improve communication and problem-solving abilities in patients and their families by sessions focused on: assessment of the individual's and the family's strengths, weaknesses, and goals; education about schizophrenia and treatment; communication skills training; problem-solving training; and special problems (Falloon et al. 1985). Treatment sessions are provided on a weekly basis for months (1 hour for each session) (groups of about 8-9 persons - patients and caregivers).
  Other Names: Family psychoeducation
  Arms: Falloon et al. Psychoeducation Program
Behavioral: Generic Treatment — The comparator is a treatment with generic informative prospect on the disorders and with the same frequencies as the Intervention. Treatment sessions are provided on a weekly basis for 6 months (1 hour for each session) (groups of about 8-9 persons - patients and caregivers).
  Arms: Generic Treatment

SUMMARY:
Background: Psychosis in the spectrum of schizophrenia (PSS) are severe mental disorders, with a high impact on disability and participation. Poor adherence to pharmacotherapy negatively impacts on the course and outcome of PSS.

Non-adherence in these patients is 41 to 50%, and it is predictive of a higher risk of relapse and readmission up to 5-time higher than in adherent patients. Falloon et al. developed a Psychoeducation Program (FPP) aimed at improving communication and problem-solving abilities in patients and their families. Past studies reported a statistically significant reduction of the risk of relapse in patients receiving the FPP, but did not take into account effects on adherence.

Objectives: To evaluate changes in adherence to pharmacotherapy in a sample of patients diagnosed with PSS (ICD-10: F20 to F29), by comparing a group exposed to the FPP with another group exposed to a treatment with generic informative prospects on the disorders provided with same attendance frequency as the FPP (Generic Treatment - GT).

Methods: 340 patients with PSS, from 10 participating units distributed in the territory of the Italian National Health System, will be enrolled, with allocation 1:1. The sample will be randomized into an exposed group (to FPP) and an unexposed group. Adherence will be assessed on a three-monthly basis with blood levels of the primary prescribed drug by High Pressure Liquid Chromatography, with a self-report, the Medication Adherence Questionnaire, and concurrently with the administration of a 4-item interview, based on a modified version of the Adherence Interview. Survival analyses will be performed using Kaplan-Meier method, followed by Log-rank test, defining as terminal events both the start of non-adherence and/or the first relapse or readmission episode. Intention-to-treat will be applied in considering the primary and secondary outcomes. Multiple imputations will be applied to integrate missing data.

Expected results: Median prevalence of non-adherence to pharmacotherapy in patients already in contact with a psychiatric service is 47%; effect size of psychosocial treatment on various outcomes, including relapse, readmission and adherence to drug is 0.48 of the standard deviation (SD), with 95% C.I.=0.10 to 0.85. The intervention is expected to produce a change in the prevalence of non-adherence to drug in the exposed group with an effect size of 0.45 SD.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of psychosis in the spectrum of schizophrenia (ICD-10: F20 to F29); -age from 18 to 55;
* being in care for 2 years or more.

Exclusion Criteria:

* mental retardation, or any severe cognitive impairment;
* psychosis due to substance abuse or to a medical condition;
* affective psychosis;
* comorbid substance dependence;
* patient does not understand Italian language;
* pharmacotherapy with depot.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Adherence | Change from baseline in adherence to treatment at 6 months
  Adherence will be checked with a triple method of assessment: patient's self-report, patient's replies to a four-query interview, and assessment of blood levels of the prescribed drug.

SECONDARY OUTCOMES:
Psychotic symptoms | Changes from baseline in levels of psychotic symptoms at 6 months, with effects maintained at12 months and 18 months
  The occurrence of psychotic symptoms, according to the Brief psychiatric Rating Scale (BPRS) and the Positive and Negative Syndrome Scale (PANSS)
General level of psychopathology | Changes from baseline in levels of general psychopathology at 6 months, with effects maintained at 12 and 18 months
  The general level of psychopathology will be measured according to the Health of the Nation rating scale (HoNOS)
Changes in the social functioning | Changes from baseline in social functioning at 6 months, maintained at 12 and 18 months
  Social functioning will be measured according to Personal and Social Performance scale (PSP). Quality of life will be measured as well, using the WHO-Quality of Life-Short version (WHOQOL-Bref).
Readmission | Occurrence of episodes of readmission over 27 months
  An episode of readmission is any admission to a psychiatric service for the necessity of controlling symptoms, behavior or therapy. Admission to the hospital for reason of somatic illness will be not considered an episode of readmission.

CONTACTS AND LOCATIONS:
Overall Officials: donatella rita petretto, PhD eq, Principal Investigator — Department of Psychology, State University of Cagliari
Locations (8):
- Italy (8):
  - Università Degli Studi Di Urbino "Carlo Bo", Urbino, Urbino/Pesaro
  - Università Degli Studi Di Bari, Bari
  - Fatebenefratelli Irccs, Brescia
  - Azienda Universitaria Ospedaliera Cagliari, Cagliari
  - Università Degli Studi Di Cagliari, Cagliari
  - Ausl 3 Centro Molise Di Campobasso, Campobasso
  - Università Degli Studi Di Catania, Catania
  - Azienda Ospedaliera Universitaria Policlinico Martino Di Messina, Messina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Falloon IR, Boyd JL, McGill CW, Williamson M, Razani J, Moss HB, Gilderman AM, Simpson GM. Family management in the prevention of morbidity of schizophrenia. Clinical outcome of a two-year longitudinal study. Arch Gen Psychiatry. 1985 Sep;42(9):887-96. doi: 10.1001/archpsyc.1985.01790320059008. PMID 2864032
- [Background] Petretto DR, Preti A, Zuddas C, Veltro F, Rocchi MB, Sisti D, Martinelli V, Carta MG, Masala C; SPERA-S group. Study on psychoeducation enhancing results of adherence in patients with schizophrenia (SPERA-S): study protocol for a randomized controlled trial. Trials. 2013 Oct 7;14:323. doi: 10.1186/1745-6215-14-323. PMID 24099414
- [Background] Petretto DR, Lussu C, Zuddas C, Pistis I, Piras P, Preti A, et al. Meta-Review of Systematic and Meta-Analytic Reviews on Family Psychoeducation for Schizophrenia. Austin J Clin Neurol 2017; 4(2): 1107.